CLINICAL TRIAL: NCT07094646
Title: An Assessment of Hematologic Diseases Among Blood Transfusion Recipients and Donated Units at a Pediatric Regional Referral Hospital in Uganda
Brief Title: Full Assessment of Clinical Transfusion Support
Acronym: FACTS
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cincinnati Children's Hospital Medical Center (CCHMC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: FACTS
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Anemia; Blood Transfusion; Malaria Parasitaemia
Keywords: FACTS; JRRH; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried Blood Spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Wet Season - Transfusion: Those receiving a blood transfusion during the Eastern Uganda wet season.
- Dry Season - Transfusion: Those receiving a blood transfusion during the Eastern Uganda dry season.
- Wet Season - Donated: Transfusion units donated during the Eastern Uganda wet season.
- Dry Season - Donated: Transfusion units donated during the Eastern Uganda dry season.

SUMMARY:
This study looks at why some children develop very severe anemia that leads to a blood transfusion. It also checks for diseases in the blood they receive. Researchers are using small samples of dried blood (called dried blood spots) from both the children and the donated blood to find out what might be causing the anemia.

DETAILED DESCRIPTION:
This study includes children at Jinja Regional Referral Hospital (Jinja, Uganda) who need a blood transfusion, whether they are in the clinic, emergency room, or children's ward. After doctors finish the usual blood tests, a small sample of leftover blood will be saved on a special card (called a dried blood spot). The same will be done for all blood transfused during the study. These samples will be frozen and later sent to Cincinnati Children's Hospital for testing.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving a blood transfusion in Eastern Uganda at Jinja Regional Referral Hospital.

Exclusion Criteria:

* If receiving a blood transfusion, refusal or inability to sign an informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving a blood transfusion in Eastern Uganda at Jinja Regional Referral Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Frequency of Sickle Cell Anemia | At enrollment.
  How common sickle cell anemia is in children who need a blood transfusion in Eastern Uganda.

SECONDARY OUTCOMES:
Frequency of Malaria Parasitemia | At enrollment.
  How common malaria parasitemia in children needing blood transfusions in Eastern Uganda.
Frequency of Iron Deficiency | At enrollment
  How often people who get blood transfusions have low iron levels, and the iron levels in the blood that is donated and used for transfusions
Blood Group Markers | At enrollment.
  Checking to ensure safe blood matches from donated blood and people receiving blood transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Jinja Regional Referral Hospital (JRRH), Jinja, Uganda

IPD SHARING:
Plan to Share IPD: No
All samples collected will be de-identified and their collection, storage and analysis constitute no more than minimal risk activities.